CLINICAL TRIAL: NCT05471752
Title: Isolation, Characterization and Evaluation of the Potential of TissuE-resideNt cElls From Waste Musculoskeletal and Associated Connective Tissues
Acronym: TENET(L4165)
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: TENET(L4165)
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general purpose of this study is characterization of tissue-resident cells derived from different musculoskeletal and/or associated connective tissues (such as cartilage, synovial membrane, synovial fluid, bone, adipose tissue and tendons), in order to identify new strategies for the treatment of degenerative and inflammatory musculoskeletal disorders. Cells isolated from different tissue sources will be compared with each other by phenotypic and functional characterization, following culture and treatment with inflammatory elements, drugs and orthobiologics. Moreover, with the aim to assess predictive markers of therapeutic success, a correlation study of the content and properties of the cells isolated from different types of tissue with the clinical profile of the enrolled patients will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* males and females

  * 18 years old
* patients undergoing elective surgery at IRCCS Istituto Ortopedico Galeazzi among which joint surgery (including hip or knee replacement), or anterior cruciate ligament (ACL) reconstruction or rotator cuff repair

Exclusion Criteria:

* age < 18 years old
* patients unable to sign the Informed Consent
* positivity to virological test (HIV, HCV, HBV, TPHA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males and females pateints, being ≥18 years old, undergoing elective surgery at IRCCS Istituto Ortopedico Galeazzi among which joint surgery (including hip or knee replacement), or anterior cruciate ligament (ACL) reconstruction or rotator cuff repair
Sampling Method: Probability Sample
Enrollment: 742 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2027-05-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
Correlation beetween patients' age and cell yield | 5 years
  The primary outcome of the study will be to identify possible correlations between the cellular yields and patients age. The data from different tissue sources will be analyzed to assess whether the changes are tissue-specific.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy